CLINICAL TRIAL: NCT05164770
Title: A Multi-center, Prospective Clinical Study of Zanubrutinib, Rituximab and Combination Chemotherapy in Patients With Newly-diagnosed Aggressive B-cell Non-Hodgkin Lymphoma
Brief Title: Study of Zanubrutinib, Rituximab and Combination Chemotherapy in Newly-diagnosed Aggressive B-cell Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Department of Hematology, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-NHL002
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: High Grade B-Cell Lymphoma, Not Otherwise Specified; High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6 Rearrangements; Diffuse Large B Cell Lymphoma; B-cell Non Hodgkin Lymphoma; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zanubrutinib+R+chemotherapy (Experimental): Zanubrutinib+R-CHOP; Zanubrutinib+R-DA-EPOCH; Zanubrutinib+R-HD MTX
  Interventions: Drug: Zanubrutinib+R-CHOP; Zanubrutinib+R-DA-EPOCH; Zanubrutinib+R-HD MTX
- R+chemotherapy (Active Comparator): R-CHOP; R-DA-EPOCH; R-HD MTX
  Interventions: Drug: R-CHOP; R-DA-EPOCH; R-HD MTX

INTERVENTIONS:
Drug: Zanubrutinib+R-CHOP; Zanubrutinib+R-DA-EPOCH; Zanubrutinib+R-HD MTX — Zanubrutinib+R-CHOP Regimen: Zanubrutinib 160mg bid; R-CHOP: Rituximab 375mg/m2 d0, Cyclophosphamide 750mg /m2 d1, Doxorubicin 50mg /m2 or Doxorubicin liposome 30-40 mg /m2 d1, Vincristine 1.4mg /m2 or Vindesine 3mg /m2 d1, Prednisone 100mg d1-5. Every 21 days is one cycle, which can be extended to 28 days per cycle according to patients' specific tolerance to chemotherapy.
  Zanubrutinib+R-DA-EPOCH Regimen: Zanubrutinib 160mg bid; R-DA-EPOCH: Rituximab 375mg/m2 d0, Etoposide 50mg/ m2, Epirubicin 15mg/ m2, Vincristine 0.4mg/ m2, d1-4, Cyclophosphamide (CTX) 750mg/ m2 d5, Prednisone 60mg/ m2 d1-5. Every 21 days is one cycle, which can be extended to 28 days per cycle according to patients' specific tolerance to chemotherapy.
  Zanubrutinib+R-HD MTX Regimen: Zanubrutinib 160mg bid; R-HD MTX: Rituximab 375mg/m2 d0, Methotrexate 3.5g/m2 d1. Every 21 days is one cycle, which can be extended to 28 days per cycle according to patients' specific tolerance to chemotherapy.
  Arms: Zanubrutinib+R+chemotherapy
Drug: R-CHOP; R-DA-EPOCH; R-HD MTX — R-CHOP: Rituximab 375mg/m2 d0, Cyclophosphamide 750mg/m2 d1, Doxorubicin 50mg/m2 or Doxorubicin liposome 30-40 mg /m2 d1, Vincristine 1.4mg/m2 or Vindesine 3mg/m2 d1, Prednisone 100mg d1-5. Every 21 days is one cycle, which can be extended to 28 days per cycle according to patients' specific tolerance to chemotherapy.
  R-DA-EPOCH: Rituximab 375mg/m2 d0, Etoposide 50mg/m2, Epirubicin 15mg/m2, Vincristine 0.4mg/ m2, d1-4, Cyclophosphamide (CTX) 750mg/ m2 d5, Prednisone 60mg/ m2 d1-5. Every 21 days is one cycle, which can be extended to 28 days per cycle according to patients' specific tolerance to chemotherapy.
  R-HD MTX: Rituximab 375mg/m2 d0, Methotrexate 3.5g/m2 d1. Every 21 days is one cycle, which can be extended to 28 days per cycle according to patients' specific tolerance to chemotherapy.
  Arms: R+chemotherapy

SUMMARY:
Non-Hodgkin lymphoma (NHL), with high aggressiveness and mortality, is one of the top ten high-incidence tumors in the world and is among the ten most prevalent cancers worldwide with the fastest growing incidence. Although novel immunotherapies represented by anti-CD20 monoclonal antibodies and CAR-T cell therapies have significantly improved the prognosis of B-NHL patients, there are still nearly one-third of patients who are resistant to initial treatment or relapse after remission. Zanubrutinib is an oral small molecule BTK inhibitor, and has shown good efficacy and safety in multiple subtypes of B-cell lymphoma. However, the efficacy of zanubrutinib in highly aggressive B-cell lymphoma remains to be further studied

DETAILED DESCRIPTION:
Non-Hodgkin lymphoma (NHL), with high aggressiveness and mortality, is one of the top ten high-incidence tumors in the world and is among the ten most prevalent cancers worldwide with the fastest growing incidence. B-cell non-Hodgkin's lymphoma (B-NHL) is the most common type of NHL. Although novel immunotherapies represented by anti-CD20 monoclonal antibodies and CAR-T cell therapies have significantly improved the prognosis of B-NHL patients, there are still nearly one-third of patients who are resistant to initial treatment or relapse after remission.

High-grade B-cell lymphoma (HGBL)-DH/TH with MYC/BCL2 and/or BCL6 translocation, accounts for about 7-10% in DLBCL. The remission rate of conventional chemotherapy is low.(ORR:32%,CR:12%). The median OS is 12 months. The survival outcome of induction chemotherapy is improved limited compared to R-CHOP. Currently, there are a lack of effective treatments options for HGBL. How to improve curative effect needs more research.

Zanubrutinib is an oral small molecule BTK inhibitor, and has shown good efficacy and safety in multiple subtypes of B-cell lymphoma. Zanubrutinib received FDA approval for adult mantle-cell lymphoma (MCL) and small lymphocytic lymphoma/chronic lymphocytic leukemia (SLL/CLL) patients who have received at least one previous treatment on 15 Nov 2019, becoming the first US-listed Chinese innovative anti-cancer drug. However, the efficacy of zanubrutinib in highly aggressive B-cell lymphoma remains to be further studied.

Therefore, we present this study protocol to add Zanubrutinib to the first-line treatment of highly aggressive B-NHL, applying zanubrutinib combined with rituximab plus chemotherapy in the treatment of highly aggressive B-NHL compared to rituximab plus chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, gender not limited
2. Newly and histologically diagnosed aggressive B-NHL
3. Patients who have not received systematic chemotherapy or immunotherapy;
4. Patients with at least ≥1 tumor foci with a measurable maximum axis exceeding 1.5 cm;
5. Eastern cancer collaboration group(ECOG) physical status score: 0-2
6. a)Blood routine: (independent of growth factor support or transfusion within 7 days of study entry) neutrophils absolute value ≥1.5×109/L, platelets ≥75×109/L, b) Coagulation function: INR ≤2.5 times ULN, c) Blood biochemistry: total bilirubin ≤2 times ULN, AST or ALT≤2.5 times ULN d) Ccr ≥ 30 mL/min;
7. expected survival time ≥3 months;
8. Willing to take contraceptive measures during the trial period and within 1 week after the trial ends;
9. Voluntarily sign written informed consent before screening.

Exclusion Criteria:

1. Current or previous malignancy, unless radical therapy has been performed and there is no evidence of recurrence or metastasis in the past 5 years;
2. Patients scheduled for major surgery(except for examination for diagnostic purposes) within 4 weeks or participating in drug/device clinical trials;
3. Prior or concurrent indolent B-cell lymphoma transformation;
4. Uncontrolled or significant cardiovascular disease;
5. Had active bleeding within 2 months prior to screening, or was taking anticoagulant drugs, or was considered by the investigator to have a clear tendency to bleeding;
6. Stroke or intracranial hemorrhage within 6 months;
7. Subjects with clinically significant gastrointestinal abnormalities that may affect drug intake, transport or absorption (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.)
8. Active or uncontrolled HBV (HBsAg positive and HBV DNA titer positive), HCV Ab positive or HIV positive;
9. Uncontrolled, active systemic fungal, bacterial, viral, or other infections (defined as showing persistent signs/symptoms related to infection, despite the use of appropriate antibiotics or other treatments without improvement)
10. Allergies or hypersensitivity reactions to zanubrutinib, rituximab or any other component of the applicable study drug;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  per 3 and 6 cycle

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 3 years
Occurrence of adverse events and serious adverse events | 3 years
  per 3 and 6 cycle
Overall Survival (OS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, PhD, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Department of Hematology, Shandong Provincial Hospital, Jinan, Shandong, China